CLINICAL TRIAL: NCT04728724
Title: Neoadjuvant Sintilimab or Combined With Chemotherapy for Stage III Driven Gene Mutation Negative Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Immunotherapy for Stage III Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-009
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Anti-PD-1 monotherapy
  Interventions: Drug: Sintilimab
- Group B (Experimental): Anti-PD-1 plus chemotherapy
  Interventions: Drug: Sintilimab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Sintilimab — Neoadjuvant treatment stage: Sintilimab 200mg, q3w, i.v., 2-4 cycles, then receive chest CT evaluation.
  Surgery stage: the patients will receive radical surgery after the neoadjuvant treatment.
  Adjuvant treatment stage: according to the NCCN guidelines.
Drug: Chemotherapy — Neoadjuvant treatment stage: Sintilimab 200mg, q3w, i.v., 2-4 cycles; platinum-based chemotherapy (Non-squamus: Carboplatin AUC 5 + Pemetrexed 500mg/m2; Squamous: Carboplatin AUC 5 + Gemcitabine 1000mg/m2 or Paclitaxel 200mg/m2) q3w, i.v., 2-4 cycles, then receive chest CT evaluation.
  Surgery stage: the patients will receive radical surgery after the neoadjuvant treatment.
  Adjuvant treatment stage: according to the NCCN guidelines.
  Arms: Group B

SUMMARY:
This is a phase II, non-randomized, open-label, multi-center study to evaluate the efficacy of neoadjuvant Sintilimab (PD-1 antibody) or combined with chemotherapy as first-line treatment in patients with stage III non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage III confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. With the feasiblility or anticipated feasiblility after neoadjuvant therapy to receive radical surgery;
8. Patients with good function of other main organs (liver, kidney, blood system, etc.):

   * ANC count ≥1.5×10^9/L, platelet count ≥100×10^9/L，hemoglobin ≥90 g/L;
   * the international standard ratio of prothrombin time (INR) and prothrombin time (PT) < 1.5 times of upper limit of normal (ULN);
   * Partial thromboplastin time (APTT) ≤1.5×ULN;
   * Total bilirubin ≤1.5×ULN;
   * Alanine aminotransferase (ALT) aspartate aminotransferase (AST) ≤2.5×ULN, or ALT and AST ≤5×ULN in the patients with liver metastatic tumor.
9. Patients with normal lung function can tolerate surgery;
10. Without systematic metastasis (including M1a, M1b and M1c);
11. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of Sintilimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
12. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of Sintilimab (whichever is later).

Exclusion Criteria:

1. Non-squamous cell carcinoma with EGFR active mutation positive or ALK rearrangement;
2. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
3. Administration of any Chinese medicine against cancer before administration of the drug;
4. Participants with other cancer (excluding cervical carcinoma in situ, cured basal cell carcinoma, bladder epithelial tumor [including TA and tis]) within five years before the start of this study;
5. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
6. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
7. Antibiotics were used to treat the infection for 4 weeks prior to the start of the trial;
8. Participants who were systemically treated with corticosteroids (prednisone or other corticosteroids >10 mg/ day) or other immunosuppressive agents within 2 weeks prior to first administration. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of less than 10 mg/ day of prednisone are permitted;
9. Participants who are allergic to the test drug or any auxiliary materials;
10. Participants with active hepatitis B, hepatitis C or HIV;
11. The vaccine was administered within 4 weeks of the start of the trial;
12. Participants who have undergone major surgery or severe trauma in other systems within 2 months before the start of this trial;
13. Pleural effusion, pericardial effusion or ascites that are not clinically controlled and require pleural puncture or abdominal puncture drainage within 2 weeks before inclusion;
14. The patients have active pia meningioma, uncontrolled or untreated brain metastases;
15. Pregnant or lactating women;
16. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
17. Participated in another therapeutic clinical study;
18. Other factors that researchers think it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | up to 5 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy.Only patients with measurable lesions at baseline will be analyzed.
Disease-free survival (DFS) | up to 60 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Progression-free survival (PFS) | up to 60 months
  It refers to the time from the first administration of drug in this study to the disease progression or death (including any cause of death in the case of no progression) as recorded in CRF, regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Safety: frequency of severe adverse events | up to 6 months
  The frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided